CLINICAL TRIAL: NCT03628105
Title: The Effect of Cognitive Restructuring Before Exposure for Claustrophobia on Expectancy and Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirstyn L. Krause (Other)
Responsible Party: Sponsor-Investigator, Kirstyn L. Krause, Principal Investigator, Toronto Metropolitan University
Organization: Toronto Metropolitan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB 2018-161
Record Dates: First submitted 2018-07-10; First posted 2018-08-14 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: CR Before:Engaging in Cognitive Intervention Before Exposure; CR After:Engaging in Cognitive Intervention After Exposure
Keywords: Anxiety; Specific Phobia; Claustrophobia; Exposure; Cognitive therapy; Cognitive restructuring; Consolidation; Inhibitory learning; Expectancy violation; Expectancy; Exposure therapy; Anxiety disorder
MeSH Terms: conditions — Anxiety Disorders; Phobia, Specific; Claustrophobia

STUDY DESIGN:
Intervention Model Description: Participants will complete baseline pretreatment outcome measures at the first visit to the lab. All participants will watch the same psychoeducation video explaining the nature of anxiety and rationale for exposure therapy. Participants will then be randomly assigned to either the CR Before condition or the CR After condition. CR Before will complete 15 minutes of CR (Preparation) before engaging in six 5-minute exposure trials in a claustrophobic chamber, and complete the 15-minute filler task after exposure. CR After will complete the 15-minute filler task before exposure, engage in six 5-minute exposure trials in a claustrophobic chamber, and engage in 15 minutes of CR (Consolidation) after exposure. Participants will complete posttreatment outcome measures immediately following the intervention. Participants will return one month later to complete followup outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CR Before Exposure (Experimental): Participants in this arm will receive 15 minutes of CR (preparation) before engaging in exposure and will complete the 15-minute questionnaire filler task after exposure.
  Interventions: Behavioral: CR Before Exposure
- CR After Exposure (Experimental): Participants in this arm will complete the 15-minute questionnaire filler task before exposure and receive 15 minutes of CR (consolidation) after engaging in exposure.
  Interventions: Behavioral: CR After Exposure

INTERVENTIONS:
Behavioral: CR Before Exposure — Participants complete 15 minutes of CR (Preparation) using the "evidence technique" outlined in the cognitive-behavioral manual Mind Over Mood (Greenberger & Padesky, 2016). This technique involves evaluating the validity of expected feared outcomes. Next, participants complete six 5-minute exposure trials using a claustrophobic chamber and other materials (e.g., scarf, mask, handcuffs). Finally, participants complete the 15-minute self-report filler task (including questions from the MMPI-2, Butcher et al., 1989) which acts as a no-treatment comparison to CR being conducted after exposure in the other arm of the study.
  Arms: CR Before Exposure
Behavioral: CR After Exposure — Participants complete the 15-minute self-report filler task (including questions from the MMPI-2, Butcher et al., 1989) which acts as a no-treatment comparison to CR being conducted before exposure in the other arm of the study. Next, participants complete six 5-minute exposure trials using a claustrophobic chamber and other materials (e.g., scarf, mask, handcuffs). Then, participants complete 15 minutes of CR (Consolidation, Craske et al.'s, 2014) by calculating the difference between predicted and actual expected feared outcomes, and identifying identify (1) whether they believe their feared outcomes occurred (Yes/No), (2) describe how they know this to be true, and (3) reflect on what they learned about their feared outcome or expectancy through exposure.
  Arms: CR After Exposure

SUMMARY:
Whether used alone or in combination with other approaches, strategies such as cognitive restructuring (CR) and exposure are well-established treatments for anxiety. CR involves identifying and challenging thoughts, beliefs, or assumptions that maintain anxiety, and exposure involves confronting feared situations, typically in a gradual manner. Many theories have been proposed to explain why exposure is effective. One theory posits that corrective learning occurs only when expectations about the outcome of a situation are violated. Therefore, exposure is thought to be effective when the discrepancy between the expected and actual outcome is maximized. One group of researches has suggested that engaging in CR prior to exposure will prematurely reduce the discrepancy between expectancy and outcome, resulting in less inhibitory learning. As such, they recommend that CR only be conducted after exposure in order to consolidate learning about expectancy violation. This recommendation has not been experimentally studied and is in contrast to what is typically practiced clinically. CR is often introduced in therapy prior to exposure. The present study will determine whether conducting CR before exposure results in (1) greater initial reductions in expectation following CR before exposure, (2) less expectancy violation, and (3) poorer treatment gains at posttreatment and 1-month followup. Eighty-two participants with claustrophobia will be randomly assigned to receive either CR before exposure or CR after exposure. The intervention will be conducted in a single session.

DETAILED DESCRIPTION:
Inhibitory learning is the extinction of a behavioral response through repeated presentations of a conditioned stimulus (CS) in the absence of an unconditioned stimulus (US, CS-noUS). The CS first elicits a behavioral response through excitatory learning - repeated pairing with the US that naturally elicits the same behavioral response (CS-US). One way that inhibitory learning can be maximized in exposure is by violating one's expectancy about CS-US relationship, such that the individual is surprised by the outcome (e.g., CS-noUS). The purpose of the present study is to evaluate the recommendation to avoid cognitive interventions before exposure. Specifically, the aim is to discover whether cognitive interventions before exposure prematurely reduce expected feared outcome ratings, leading to smaller expectancy violation and poorer inhibitory learning (i.e., exposure session or intervention gains) compared to conducting exposures with a consolidation period following exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported proficiency in English language.
2. High claustrophobic fear as demonstrated by:

   1. Self-report of moderate anxiety (score of at least 2 out of 4) if participant had to lie down in small dark chamber without windows for several minutes.
   2. Endorsement of claustrophobia according to the DSM-5 criteria for Specific Phobia, with or without Criterion F.
   3. Exiting of wooden claustrophobic chamber before 2 minutes have passed, or self-reported fear rating at or exceeding 50/100 fear while in the chamber.

Exclusion Criteria:

1. Current or past cognitive behavioral therapy (i.e., cognitive therapy, exposure) for claustrophobia or anxiety and related disorders in the past year
2. Change in dose of psychotropic medication in the past 3 months.
3. Use of benzodiazepine more frequently than once per week in the past 3 months.
4. Diagnosis of current (past month) panic disorder or agoraphobia.
5. Claustrophobia due to or worsened by current (past month) posttraumatic stress disorder (PTSD).
6. Participants with current (past month) diagnosis of severe depression, bipolar disorder, alcohol/substance use, or psychosis.
7. Presence of imminent suicidality or homicidality.
8. Self-reported medical condition that may make it dangerous for participant to experience heightened emotions or arousal (e.g., heart condition/disease, respiratory problem, asthma triggered by intense emotion/arousal).
9. Participation in professional treatment for claustrophobia between the end of the first lab meeting and the 1-month follow-up (Note: This does not include self-help exposure practice).
10. Weight or height exceeding maximum capacity of claustrophobic chamber (e.g., weight over 250 lbs, height over 6 feet 5 inches).

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Change from pretreatment (i.e., baseline) Behavioral Approach Test (BAT): Behavioral Approach at posttreatment and 1-month follow-up | Administered before the intervention on day 1 (pretreatment), immediately after the intervention on day 1 (posttreatment, same day as pretreatment) and at 1-month follow-up.
  The BAT includes eight 30-second cumulative steps designed to elicit increasing fear of suffocation and restriction (e.g., sleeping bag, mask, hand-cuffs, blankets), and is adapted from Deacon et al. (2010). An index of behavioral approach will be calculated by summing the number of points accrued in each step.
Change from pretreatment (i.e., baseline) Behavioral Approach Test (BAT): Peak Fear at posttreatment and 1-month follow-up | Administered before the intervention on day 1 (pretreatment), immediately after the intervention on day 1 (posttreatment, same day as pretreatment) and at 1-month follow-up.
  Self-report measure assessing the highest level of fear experienced during the final completed step of the BAT at pretreatment from 0% (No Fear) to 100% (Extreme fear).
Change from pretreatment (i.e., baseline) self-reported claustrophobic anxiety as measured by Claustrophobia Questionnaire: Total score at posttreatment and 1-month follow-up | Administered before the intervention on day 1 (pretreatment), immediately after the intervention on day 1 (posttreatment, same day as pretreatment) and at 1-month follow-up.
  Self-report measure assessing the severity of claustrophobic anxiety in situations eliciting fear of suffocation and restriction. 26 items are summed to create a total score. Total scores range from 0 to 104 with higher scores indicating greater claustrophobic anxiety.

SECONDARY OUTCOMES:
Behavioral Approach Test (BAT): Urge to Escape | Administered before the intervention on day 1 (pretreatment), immediately after the intervention on day 1 (posttreatment, same day as pretreatment) and at 1-month follow-up.
  Self-report measure assessing the strongest urge to escape experienced during the final completed step of the BAT at pretreatment from 0% (No Urge to Escape) to 100% (Extreme Urge to Escape).
Self-reported Suffocation Anxiety as measured by the Claustrophobia Questionnaire: Suffocation subscale | Administered before the intervention on day 1 (pretreatment), immediately after the intervention on day 1 (posttreatment, same day as pretreatment) and at 1-month follow-up.
  Subscale self-report measure assessing the severity of claustrophobic anxiety in situations eliciting fear of suffocation. Fourteen items are summed to create a subscale score. Scores range from 0 to 56 with greater scores indicating greater suffocation anxiety.
Self-reported Restriction Anxiety as measured by the Claustrophobia Questionnaire: Restriction subscale | Administered before the intervention on day 1 (pretreatment), immediately after the intervention on day 1 (posttreatment, same day as pretreatment) and at 1-month follow-up.
  Subscale self-report measure assessing the severity of claustrophobic anxiety in situations eliciting fear of restriction. Twelve items are summed to create a subscale score. Scores range from 0 to 48 with greater scores indicating greater restriction anxiety.
Self-reported Fear of Suffocation as measured by the Claustrophobia General Cognitions Questionnaire: Suffocation subscale | Administered before the intervention on day 1 (pretreatment), immediately after the intervention on day 1 (posttreatment, same day as pretreatment) and at 1-month follow-up.
  Subscale self-report measure of the likelihood of claustrophobic cognitions about suffocation while in enclosed spaces. Eight items are summed to create a subscale score. Scores range from 0 to 40 with greater scores indicating greater fear of suffocation.
Self-reported Fear of Inability to Escape as measured by the Claustrophobia General Cognitions Questionnaire: Inability to Escape subscale | Administered before the intervention on day 1 (pretreatment), immediately after the intervention on day 1 (posttreatment, same day as pretreatment) and at 1-month follow-up.
  Subscale self-report measure of the likelihood of claustrophobic cognitions about inability to escape while in enclosed spaces. Eight items are summed to create a subscale score. Scores range from 0 to 40 with greater scores indicating greater fear of inability to escape.
Self-reported Fear of Loss of Control as measured by the Claustrophobia General Cognitions Questionnaire: Loss of control subscale | Administered before the intervention on day 1 (pretreatment), immediately after the intervention on day 1 (posttreatment, same day as pretreatment) and at 1-month follow-up.
  Subscale self-report measure of the likelihood of claustrophobic cognitions about loss of control while in enclosed spaces. Nine items are summed to create a subscale scores. Scores range from 0 to 45 with greater scores indicating greater fear of loss of control.
Expected Feared Outcome: Personal | Administered eight times on day 1 (during the intervention) and one time at 1-month follow-up.
  Verbal self-report measure evaluating the extent to which the participant believes his or her personal expected feared (selected from the CGCQ) would occur in a frightening claustrophobic exposure exercise for a specified duration on a scale from 0% (Not at all) to 100% (Completely).
Expected Feared Outcome: Suffocation | Administered eight times on day 1 (during the intervention) and one time at 1-month follow-up.
  Verbal self-report measure used to evaluate the extent to which the participant believes he or she will suffocate when in a frightening claustrophobic exposure exercise for a specified duration on a scale from 0% (Not at all) to 100% (Completely).
Expected Feared Outcome: Restriction | Administered eight times on day 1 (during the intervention) and one time at 1-month follow-up.
  Verbal self-report measure used to evaluate the extent to which the participant believes he or she will become trapped when in a frightening claustrophobic exposure exercise for a specified duration on a scale from 0% (Not at all) to 100% (Completely).
Expected Feared Outcome: Peak Fear | Administered eight times on day 1 (during the intervention) and one time at 1-month follow-up.
  Verbal self-report measure used to evaluate the highest amount of fear participants believe they will experience in a frightening claustrophobic exposure exercise for a specified duration on a scale from 0% (No Fear) to 100% (Extreme Fear).
Expected Feared Outcome: Urge to Escape | Administered eight times on day 1 (during the intervention) and one time at 1-month follow-up.
  Verbal self-report measure used to evaluate the strongest urge to escape participants believe they will experience in a frightening claustrophobic exposure exercise for a specified duration on a scale from 0% (No Urge to Escape) to 100% (Extreme Urge to Escape).
Perceived Actual Outcome: Peak Fear | Administered six times on day 1 (during the intervention) and one time at 1-month follow-up.
  The highest level of fear the participant experienced during the previous claustrophobic exposure trial on a scale from 0% (No Fear) to 100% (Extreme fear).
Perceived Actual Outcome: Urge to Escape | Administered six times on day 1 (during the intervention) and one time at 1-month follow-up.
  The strongest urge to escape the participant experienced during the previous claustrophobic exposure trial on a scale from 0% (No urge to escape) to 100% (Extreme urge to escape).
Mean Expectancy Violation: Personal | Mean of 6 Expectancy Violation: Personal change scores calculated on day 1 during the intervention.
  The mean of the 6 change scores calculated for Expectancy Violation: Personal (i.e., the difference between the Perceived Actual Outcome: Personal rating after each exposure trial from the Expected Feared Outcome: Personal rating before each exposure trial - see Other pre-specified outcomes). Scores can range between 0% and 100% with greater scores indicating greater Mean Expectancy Violation: Personal.
Mean Expectancy Violation: Suffocation | Mean of 6 Expectancy Violation: Suffocation change scores calculated on day 1 during the intervention.
  The mean of the 6 change scores calculated for Expectancy Violation: Suffocation (i.e., the difference between the Perceived Actual Outcome: Suffocation rating after each exposure trial from the Expected Feared Outcome: Suffocation rating before each exposure trial - see Other pre-specified outcomes). Scores can range between 0% and 100% with greater scores indicating greater Mean Expectancy Violation: Suffocation.
Mean Expectancy Violation: Restriction | Mean of 6 Expectancy Violation: Restriction change scores calculated on day 1 during the intervention.
  The mean of the 6 change scores calculated for Expectancy Violation: Restriction (i.e., the difference between the Perceived Actual Outcome: Restriction rating after each exposure trial from the Expected Feared Outcome: Restriction rating before each exposure trial - see Other pre-specified outcomes). Scores can range between 0% and 100% with greater scores indicating greater Mean Expectancy Violation: Restriction.

OTHER OUTCOMES:
Self-reported depression, anxiety, and stress as measured by the Depression Anxiety Stress Scales (21-item version) | Administered once on day 1 at pretreatment.
  Self-report questionnaire measuring emotional states of depression, anxiety, and stress in the past week. Each subscale contains 7 items, which are first summed, then doubled. Scores on each subscale can range from 0 to 42, with greater scores indicating greater levels of distress
Treatment expectancy and credibility as measured by the Credibility/Expectancy Questionnaire | Administered once on day 1 during the intervention.
  Self-report measure assessing the perceived credibility and expectancy of exposure therapy. Answers to each of the 6 items are transformed into standard scores and summed to create either a total score, or a subscale credibility score or treatment expectancy score. The range of scores is not exact given that standard scores indicate deviations from the mean. According to the normal distribution, approximately 99.7% of participants should fall within a score -3 and +3 for each item, yielding a likely total range between -15 and +15 for the total score and -9 and +9 for each subscale score (credibility, treatment expectancy). Greater scores indicating greater treatment expectancy and credibility ratings.
Perceived Actual Outcome: Personal | Administered six times on day 1 (during the intervention) and one time at 1-month follow-up.
  Verbal self-report measure used to evaluate how strongly the participant believes their Expected Feared Outcome: Personal actually occurred during the previous claustrophobic exposure trial on a scale from 0% (Not at all) to 100% (Completely).
Perceived Actual Outcome: Suffocation | Administered six times on day 1 (during the intervention) and one time at 1-month follow-up.
  Verbal self-report measure used to evaluate how strongly the participant believes their Expected Feared Outcome: Suffocation actually occurred during the previous claustrophobic exposure trial on a scale from 0% (Not at all) to 100% (Completely).
Perceived Actual Outcome: Restriction | Administered six times on day 1 (during the intervention) and one time at 1-month follow-up.
  Verbal self-report measure used to evaluate how strongly the participant believes their Expected Feared Outcome: Restriction actually occurred during the previous claustrophobic exposure trial on a scale from 0% (Not at all) to 100% (Completely).
Expectancy Violation: Personal | Change score calculated using expected feared outcome and perceived actual outcome ratings completed 6 times (for each of the 6 exposure trials) on day 1 during the intervention.
  Change score calculated by subtracting the Perceived Actual Outcome: Personal rating (see "Other Pre-specified Outcome Measures" for definition) after each exposure trial from the Expected Feared Outcome: Personal rating before each exposure trial. Scores can range between 0% and 100% with greater scores indicating greater Expectancy Violation: Personal.
Expectancy Violation: Suffocation | Change score calculated using expected feared outcome and perceived actual outcome ratings completed 6 times (for each of the 6 exposure trials) on day 1 during the intervention.
  Change score calculated by subtracting the Perceived Actual Outcome: Suffocation rating (see "Other Pre-specified Outcome Measures" for definition) after each exposure trial from the Expected Feared Outcome: Suffocation rating before each exposure trial. Scores can range between 0% and 100% with greater scores indicating greater Expectancy Violation: Suffocation.
Expectancy Violation: Restriction | Change score calculated using expected feared outcome and perceived actual outcome ratings completed 6 times (for each of the 6 exposure trials) on day 1 during the intervention.
  Change score calculated by subtracting the Perceived Actual Outcome: Restriction rating (see "Other Pre-specified Outcome Measures" for definition) after each exposure trial from the Expected Feared Outcome: Restriction rating before each exposure trial. Scores can range between 0% and 100% with greater scores indicating greater Mean Expectancy Violation: Suffocation.

CONTACTS AND LOCATIONS:
Overall Officials: Kirstyn L Krause, MA, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Results of the study will be disseminated via conference presentations, journal publications, and through the investigator's lab website. Upon request, de-identified aggregate participant data may be made available to a publishing journal or individual research group. Individual research groups interested in accessing de-identified data will be required to submit a proposal detailing their intended use of the data. Their qualifications will be reviewed based on their proposal and CVs. Individual research groups approved for access will be required to agree to not attempt to re-identify participants, not further distribute data, and not use the data for purposes other than specified in their original proposal. No individual data will be shared.

REFERENCES:
- [Background] Craske MG, Kircanski K, Zelikowsky M, Mystkowski J, Chowdhury N, Baker A. Optimizing inhibitory learning during exposure therapy. Behav Res Ther. 2008 Jan;46(1):5-27. doi: 10.1016/j.brat.2007.10.003. Epub 2007 Oct 7. PMID 18005936
- [Background] Craske MG, Treanor M, Conway CC, Zbozinek T, Vervliet B. Maximizing exposure therapy: an inhibitory learning approach. Behav Res Ther. 2014 Jul;58:10-23. doi: 10.1016/j.brat.2014.04.006. Epub 2014 May 9. PMID 24864005
- [Background] Deacon BJ, Sy JT, Lickel JJ, Nelson EA. Does the judicious use of safety behaviors improve the efficacy and acceptability of exposure therapy for claustrophobic fear? J Behav Ther Exp Psychiatry. 2010 Mar;41(1):71-80. doi: 10.1016/j.jbtep.2009.10.004. Epub 2009 Oct 24. PMID 19892318
- [Derived] Krause KL, Koerner N, Antony MM. Cognitive Restructuring Before Versus After Exposure: Effect on Expectancy and Outcome in Individuals With Claustrophobia. Behav Modif. 2022 Nov;46(6):1432-1459. doi: 10.1177/01454455221075754. Epub 2022 Feb 12. PMID 35156404